CLINICAL TRIAL: NCT01401036
Title: Clinical Trial of Nobori Versus Uncoated Stents In Acute Myocardial Infarction
Brief Title: Nobori And Uncoated Stent In Coronary Attack
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient data collection
Sponsor: Shigeru Saito (Network)
Collaborators: NPO International TRI Network (Network)
Responsible Party: Sponsor-Investigator, Shigeru Saito, Director, Cardiology, Shonan Kamakura General Hospital, NAUSICA Investigators
Organization: NAUSICA Investigators (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110629
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Acute Myocardial Infarction
Keywords: acute myocardial infarction; stents; angioplasty; thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nobori (Active Comparator): subjects receiving Biolimus A9 eluting stent implantation
  Interventions: Device: Biolimus A9 eluting stents
- Uncoated stents (Sham Comparator): subjects receiving uncoated stent implantation
  Interventions: Procedure: uncoated stent

INTERVENTIONS:
Device: Biolimus A9 eluting stents — implantation of Biolimus A9 eluting stents
  Other Names: Nobori® Drug Eluting Stent made by Terumo Corporation
  Arms: Nobori
Procedure: uncoated stent — implantation of any uncoated bare metal stents currently available in Japan
  Arms: Uncoated stents

SUMMARY:
Drug-eluting stents reduce rates of restenosis and reintervention, as compared with uncoated stents. Data are limited regarding the safety and efficacy of Nobori (Biolimus A9 Eluting Stent) in primary percutaneous coronary intervention (PCI) for acute myocardial infarction (AMI). Accordingly, the investigators will compare the outcomes of primary PCI for AMI between patients receiving Nobori versus uncoated stents.

ELIGIBILITY:
Inclusion Criteria:

* age more than 20 years old
* chest pain lasting more than 20 min
* symptoms beginning within 12 hours before characterization
* electrocardiogram showing ST-segment elevation or new appearance of left bundle branch block
* increase in cardiac enzymes to more than 5-fold the normal laboratory values
* infarct-related vessel are anatomically suitable for percutaneous revascularization
* patients gave their signed, informed consent

Exclusion Criteria:

* previous stent implantation within 30 days
* allergy to any of the followings : aspirin, heparin, clopidogrel, biolimus A9 or its derivatives, stainless steel 316L, PLA (Poly-Lactic Acid) Polymer or its derivatives, and contrast media
* elective surgery scheduled within 6 months
* renal insufficiency with creatinine level of more than 2.5 mg/dL
* patients associated with bleeding and/or clotting disorders, and those refusing blood transfusion
* history of massive gastrointestinal or urinary tract bleeding within 6 months
* patients currently enrolled in other clinical trials
* pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1537 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2015-08-05 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
major adverse cardiac and cerebrovascular events (MACE) | 1 year
  MACE includes all-cause death, myocardial infarction, cerebrovascular events, and target lesion revascularization

SECONDARY OUTCOMES:
major adverse cardiac and cerebrovascular events (MACE) | 1 week
  MACE includes all-cause death, myocardial infarction, cerebrovascular events, and target lesion revascularization
stent thrombosis | 1 week and 1 year
target lesion revascularization | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Saito, MD, Principal Investigator — NPO International TRI Network
Locations (50):
- Japan (50):
  - Shonan Atsugi Hospital, Atsugi, Kanagawa
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Tokyo nishi tokusyukai hospital, Akishima
  - Shonan Atsugi hospital, Atsugi
  - Tokai University Hachioji Hospital, Hachiōji
  - Hakodate Municipal Hospital, Hakodate
  - Hiratsuka kyosai hospital, Hiratsuka
  - Tokai University Hospital, Isehara
  - Ishikawa Prefectural Central Hospital, Ishikawa
  - Kanazawa Cardiovascular Hospital, Kanazawa
  - Kasukabe chuo general Hospital, Kasukabe
  - St.Marianna University School of Medicine Hospital, Kawasaki
  - Chikamori Hospital, Kochi
  - Komaki Municipal Hospital, Komaki
  - Saitama Tobu Junkanki Hospital, Koshigoe
  - Kurashiki Sentral Hospital, Kurashiki
  - Kyoto Katsura Hospital, Kyoto
  - Hayama Heart Center, Miura
  - Omuta Tenryo Hospital, Omuta
  - Osaki citizen hospital, Ōsaki
  - Saga Medical University Hospital, Saga
  - Saga-ken Medical Center Koseikan, Saga
  - Toshiba Rinkan Hospital, Sagamihara
  - Hokkaido Syakaihoken Hospital, Sapporo
  - Sapporo Hogashi Tokusyukai Hospital, Sapporo
  - Sapporo Tokusyukai Hospital, Sapporo
  - Sasebo Chuo hospital, Sasebo
  - Tosei General Hospital, Seto
  - Jichi Medical University Hospital, Shimotsuke
  - Sakurakai Takahashi Hospital, Suma
  - Taoka Hospital, Tokushima
  - Tokushima medical university hospital, Tokushima
  - Imus Katsushika Heart Center, Tokyo
  - Showa University Fujigaoka Hospital, Tokyo
  - Showa University Hospital, Tokyo
  - The Cardiovascular Institute, Tokyo
  - Toho University Hospital, Tokyo
  - Toho university ohashi medical center, Tokyo
  - Tokyo Medical and Dental Universtity Hospital, Tokyo
  - Tokyo medical University hospital, Tokyo
  - Toyama Prefectural Central Hospital, Toyama
  - Izumikawa Hospital, Unzen
  - Urazoe general hospital, Urazoe
  - Shonai Amarume Hospital, Yamagata
  - Saiseikai Yamaguchi General Hospital, Yamaguchi
  - Yamato Seiwa Hospital, Yamato
  - Yao General Hospital, Yao
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
  - Saiseikai Yokohama Tobu Hospital, Yokohama
  - Yokohama Medical University Hospital, Yokohama